CLINICAL TRIAL: NCT02766556
Title: The Effect of Dexamedetomidine for Interscalene Brachial Plexus Block on Plasma Cortisol and IL-6 After Rotator Cuff Repair: a Prospective Randomized Study
Brief Title: The Effect of Dexamedetomidine for Interscalene Brachial Plexus Block on Plasma Biomarkers After Rotator Cuff Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jae Jun Lee, associate professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2013-112
Record Dates: First submitted 2016-05-03; First posted 2016-05-10 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Saline Solution; Analgesia; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- arm 1 (Active Comparator): received ISB with 8mL of ropivacaine with 100 μg (1ml) of dexmedetomidine
  Interventions: Drug: dexmedetomidine; Procedure: ISB; Drug: Ropivacaine
- arm 2 (Placebo Comparator): received ISB with 8mL of ropivacaine with 1ml of normal saline
  Interventions: Procedure: ISB; Drug: Ropivacaine

INTERVENTIONS:
Drug: dexmedetomidine — ISB with ropivacaine with dexmedetomidine or normal saline
  Other Names: dexmedetomidine or normal saline
  Arms: arm 1
Procedure: ISB — ISB with ropivacaine with dexmedetomidine or normal saline
  Other Names: ISB for pain control
Drug: Ropivacaine — ISB with ropivacaine with dexmedetomidine or normal saline
  Other Names: ISB using ropivacaine

SUMMARY:
The present study was designed to test the hypothesis that dexmedetomidine added to ropivacaine for interscalene brachial plexus blocks for elective shoulder surgery would enhance the duration and effect of analgesia when compared with ropivacaine alone, and their influence on serum IL-6, cortisol, IL-1beta, IL-8, and substance p.

DETAILED DESCRIPTION:
Background The incidence of severe postoperative pain after shoulder surgery is 30% to 70%.The postoperative pain should be relieved for early rehabilitation and recovery. Patient-controlled analgesia (PCA) with opiate therapy may control some of the postoperative pain, but it has several side effects such as nausea, vomiting, and dizziness, which can prevent early discharge. Conversely, there are several regional blocks to control postoperative pain. Interscalene brachial plexus block (ISB) is known as one of the most effective regional blocks for shoulder surgery, but it has relatively short duration of effect.

Dexmedetomidine (DEX), a selective agonist of α2-adrenergic receptors, can be an effective adjuvant to local anesthetics for peripheral nerve block. Preclinical and clinical studies have described prolonged duration of analgesia when dexmedetomidine was added to bupivacaine, levobupivacaine, or ropivacaine for peripheral perineural blocks.

Pro-inflammatory cytokines, such as interleukin-6 (IL-6), shows a high association with acute pain because they sensitize the nervous system. IL-6 levels in the plasma are detectable 60 minutes after injury, peaking at 4-6 hours, and are proportional to tissue injury.

Increased plasma cortisol concentrations can be detected within 15 minutes following exposure to a stressor. And several biomarkers related to pain have been studying.

Method 50 patients with rotator cuff tears who had undergone arthroscopic rotator cuff repairs were enrolled in this study. Rotator cuff tears were diagnosed by preoperative magnetic resonance imaging, and the size of the rotator cuff was confirmed at the time of arthroscopic operation. Indication for surgery was a symptomatic full-thickness rotator cuff tear or a partial thickness rotator cuff tear of more than 50% thickness in case of failed conservative therapy. Twenty-five patients were randomly allocated to group 1 and received both ISB with 8mL of ropivacaine with 100 μg (1ml) of dexmedetomidine . The other 25 patients were allocated to group 2 and received ISB with 8mL of ropivacaine with 1ml of normal saline.

Power analysis indicated that a total sample size of 46 patients (23 patients in each cohort) would provide a statistical power of 99% with a 2-sided a level of 0.05 to detect significant differences in the visual analog scale (VAS) score at 6 hours postoperatively, assuming an effect size of 0.88 (mean difference, 2.46, standard deviation, 2.8). This was based on the mean and standard deviation of the VAS at 6 hours postoperatively observed in a pilot study of 20 patients.

Double-blinded randomization was performed as follows. The remaining 50 patients were randomly assigned to 1 of 2 groups depending on the additional dexmedetomidine. Randomization was performed with a computerized random-sequence generator by an independent nurse who prepared a syringe for added dexmedetomidine or saline according to the assignment. The patients and all the medical staff who participated in the operation were blinded of the assignment.

VAS pain score, IL-6, cortisol, IL-1beta, IL-8, and substance p, height, and weight were checked preoperatively. All ISB were performed preemptively under ultrasonographic guidance. After sterile preparation and draping of the injection area, the structures of the brachial plexus were identified using ultrasound (Sonosite M-Turbo 13 mHz linear probe; Sonosite Corp, Bothell, Washington). Injections were performed using an out-of-plane technique using a plexus needle (Plexus Nano Line Uniplex, 22 gauge, 50 mm; Pajunk Corp, Geisingen, Germany). Nerve stimulation was not conducted.

PCA was set at a fixed dose (fentanyl, 0.05 mg/kg loading dose and 0.03 mg/min/kg continuous dose) to remove the effect of a variable amount of PCA. VAS pain score, IL-6, cortisol, IL-1beta, IL-8, and substance p, were checked 1, 6, 12, 24, and 48 hours postoperatively. VAS pain score was selected from 0 to 10, with 0 being no pain and 10 being the most severe pain that the patient had ever experienced.

ELIGIBILITY:
Inclusion Criteria:

1. a definite rotator cuff tear that needed repair seen on preoperative magnetic resonance imaging
2. acceptance of arthroscopic surgery including rotator cuff repair
3. age more than 20 years,
4. acceptance of preemptive regional block , PCA and blood sampling after 1 ,6, 12, 24, 48 hour postoperatively. .

Exclusion Criteria:

1. they did not undergo arthroscopic rotator cuff repair
2. they stopped PCA before 48 hours postoperatively because of associated side effects
3. there was a history of a previous shoulder operation or fracture
4. there was a concomitant neurologic disorder around the shoulder
5. refusal of blood sampling.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
change of five biomarkers (IL-6 in pg/ml, cortisol in ng/ml, IL-8 in pg/ml, IL-1beta in pg/ml, substance p in pg/ml) level due to pain after shoulder surgery. | change from preoperation(baseline) IL-6, cortisol, IL-8, IL-1beta, and substance p level 1, 6, 12, 24, 48 hours after surgery due to postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: Jae Jun Lee, M.D., Principal Investigator — Department of Anesthesiology and Pain medicine, Chuncheon Sacred Heart Hospital, College of Medicine, Hallym University

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Lee SM, Park SE, Nam YS, Han SH, Lee KJ, Kwon MJ, Ji JH, Choi SK, Park JS. Analgesic effectiveness of nerve block in shoulder arthroscopy: comparison between interscalene, suprascapular and axillary nerve blocks. Knee Surg Sports Traumatol Arthrosc. 2012 Dec;20(12):2573-8. doi: 10.1007/s00167-012-1950-5. Epub 2012 Mar 21. PMID 22434159
- [Result] Moote CA. The prevention of postoperative pain. Can J Anaesth. 1994 Jun;41(6):527-33. doi: 10.1007/BF03011550. PMID 7915209
- [Result] Fritsch G, Danninger T, Allerberger K, Tsodikov A, Felder TK, Kapeller M, Gerner P, Brummett CM. Dexmedetomidine added to ropivacaine extends the duration of interscalene brachial plexus blocks for elective shoulder surgery when compared with ropivacaine alone: a single-center, prospective, triple-blind, randomized controlled trial. Reg Anesth Pain Med. 2014 Jan-Feb;39(1):37-47. doi: 10.1097/AAP.0000000000000033. PMID 24317234
- [Result] Brummett CM, Norat MA, Palmisano JM, Lydic R. Perineural administration of dexmedetomidine in combination with bupivacaine enhances sensory and motor blockade in sciatic nerve block without inducing neurotoxicity in rat. Anesthesiology. 2008 Sep;109(3):502-11. doi: 10.1097/ALN.0b013e318182c26b. PMID 18719449
- [Result] Brummett CM, Amodeo FS, Janda AM, Padda AK, Lydic R. Perineural dexmedetomidine provides an increased duration of analgesia to a thermal stimulus when compared with a systemic control in a rat sciatic nerve block. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):427-31. doi: 10.1097/AAP.0b013e3181ef4cf0. PMID 20814283
- [Result] Brummett CM, Padda AK, Amodeo FS, Welch KB, Lydic R. Perineural dexmedetomidine added to ropivacaine causes a dose-dependent increase in the duration of thermal antinociception in sciatic nerve block in rat. Anesthesiology. 2009 Nov;111(5):1111-9. doi: 10.1097/ALN.0b013e3181bbcc26. PMID 19858875
- [Result] Esmaoglu A, Yegenoglu F, Akin A, Turk CY. Dexmedetomidine added to levobupivacaine prolongs axillary brachial plexus block. Anesth Analg. 2010 Dec;111(6):1548-51. doi: 10.1213/ANE.0b013e3181fa3095. Epub 2010 Oct 1. PMID 20889939
- [Result] Marhofer D, Kettner SC, Marhofer P, Pils S, Weber M, Zeitlinger M. Dexmedetomidine as an adjuvant to ropivacaine prolongs peripheral nerve block: a volunteer study. Br J Anaesth. 2013 Mar;110(3):438-42. doi: 10.1093/bja/aes400. Epub 2012 Nov 15. PMID 23161360
- [Result] Obayah GM, Refaie A, Aboushanab O, Ibraheem N, Abdelazees M. Addition of dexmedetomidine to bupivacaine for greater palatine nerve block prolongs postoperative analgesia after cleft palate repair. Eur J Anaesthesiol. 2010 Mar;27(3):280-4. doi: 10.1097/EJA.0b013e3283347c15. PMID 19935071
- [Result] Swami SS, Keniya VM, Ladi SD, Rao R. Comparison of dexmedetomidine and clonidine (alpha2 agonist drugs) as an adjuvant to local anaesthesia in supraclavicular brachial plexus block: A randomised double-blind prospective study. Indian J Anaesth. 2012 May;56(3):243-9. doi: 10.4103/0019-5049.98767. PMID 22923822
- [Result] Brummett CM, Hong EK, Janda AM, Amodeo FS, Lydic R. Perineural dexmedetomidine added to ropivacaine for sciatic nerve block in rats prolongs the duration of analgesia by blocking the hyperpolarization-activated cation current. Anesthesiology. 2011 Oct;115(4):836-43. doi: 10.1097/ALN.0b013e318221fcc9. PMID 21666435
- [Result] Brenn D, Richter F, Schaible HG. Sensitization of unmyelinated sensory fibers of the joint nerve to mechanical stimuli by interleukin-6 in the rat: an inflammatory mechanism of joint pain. Arthritis Rheum. 2007 Jan;56(1):351-9. doi: 10.1002/art.22282. PMID 17195239
- [Result] Buenaver LF, Edwards RR, Smith MT, Gramling SE, Haythornthwaite JA. Catastrophizing and pain-coping in young adults: associations with depressive symptoms and headache pain. J Pain. 2008 Apr;9(4):311-9. doi: 10.1016/j.jpain.2007.11.005. Epub 2007 Dec 31. PMID 18165160
- [Result] Buvanendran A, Kroin JS, Berger RA, Hallab NJ, Saha C, Negrescu C, Moric M, Caicedo MS, Tuman KJ. Upregulation of prostaglandin E2 and interleukins in the central nervous system and peripheral tissue during and after surgery in humans. Anesthesiology. 2006 Mar;104(3):403-10. doi: 10.1097/00000542-200603000-00005. PMID 16508385
- [Result] Frank LA, Kunkle GA, Beale KM. Comparison of serum cortisol concentration before and after intradermal testing in sedated and nonsedated dogs. J Am Vet Med Assoc. 1992 Feb 15;200(4):507-10. PMID 1559888
- [Derived] Hwang JT, Jang JS, Lee JJ, Song DK, Lee HN, Kim DY, Lee SS, Hwang SM, Kim YB, Lee S. Dexmedetomidine combined with interscalene brachial plexus block has a synergistic effect on relieving postoperative pain after arthroscopic rotator cuff repair. Knee Surg Sports Traumatol Arthrosc. 2020 Jul;28(7):2343-2353. doi: 10.1007/s00167-019-05799-3. Epub 2019 Nov 26. PMID 31773201